CLINICAL TRIAL: NCT05929612
Title: A Phase II Study of Response Adapted Ultra Low Dose 4 Gy Radiation for Definitive Therapy of Marginal Zone Lymphoma
Brief Title: A Study of Response Adapted Ultra Low Dose 4 Gy Radiation for Definitive Therapy of Marginal Zone Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0237; NCI-2023-05151 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-06-26; First posted 2023-07-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultra Low Dose 4 Gy Radiation (Experimental): Participants will receive the ultra-low doses of radiation therapy over 1-2 days
  Interventions: Radiation: Ultra Low Dose 4 Gy Radiation

INTERVENTIONS:
Radiation: Ultra Low Dose 4 Gy Radiation — 4 Gy in 2 fractions

SUMMARY:
To learn if response-adapted, ultra-low dose radiation therapy can help to control MZL. This means participates first receive lower does of radiation therapy and then, based on how the disease responds, may receive higher doses after that.

DETAILED DESCRIPTION:
Primary Objectives:

--To evaluate the efficacy of response adapted ultra low dose therapy (4 Gy with additional 12 Gy if needed) as a complete response after completion of the program

Secondary Objectives:

* To evaluate distant recurrence of marginal zone lymphoma at 24 months
* To evaluate in field relapse at 24 months for all patients
* To evaluate the efficacy of response adapted ultra low dose therapy (4 Gy with additional 12 Gy if needed) as overall response rate (ORR) after completion of the program
* To evaluate overall survival of patients included in the study

Exploratory Objectives:

* To determine if microbiome assessment can predict response to ultra low dose radiation therapy and evaluate the differences in patient microbiome for patients who respond well and poorly to low dose radiation.
* To encourage optional co-enrollment on study PA18-0644 to facilitate collection and archiving of blood-based biomarkers and microbiome samples for patients receiving ultra low dose radiation therapy.
* To evaluate PETCT-based features for any patients receive PETCT for initial and follow up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older. Because no RT dosing data are currently available on the use of response adapted ultra low dose RT in patients <18 years of age, children are excluded from this study.
* Patients with stage I-II marginal zone lymphoma. Patients with a pathology report consistent with low grade B cell lymphoma, favor marginal zone lymphoma, are included. Other low grade lymphomas including follicular grade I/II and chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) are ineligible.
* Patients should not be planned for any systemic therapy before the first follow up evaluation after radiation (intent is to treat with radiation therapy alone).
* Patients with biopsy-proven disease treated with another modality (such as systemic therapy) prior to radiation must have clinical or radiographic evidence of residual disease before enrollment. Patients with clinical and/or radiographic masses that are measurable will have dimensions noted prior to therapy. If an excisional biopsy is performed, patients should have clinically or radiographically apparent disease after biopsy (this does not apply to gastric MALT lymphoma patients).
* Prior systemic therapy is allowed, as long as administration is prior to most recent disease assessment by imaging, clinical exam, or endoscopy. There are no limits on the nature or amount of prior systemic therapy.
* Prior antibiotics intended to treat marginal zone lymphoma are allowed, as long as administration is prior to most recent disease assessment by imaging, clinical exam, or endoscopy.
* Prior topical therapies (e.g. steroid) intended to treat cutaneous lymphoma are allowed, as long as administration is prior to most recent disease assessment by imaging, clinical exam, or endoscopy.
* For patients with gastric MALT lymphoma, H. pylori testing by immunohistochemistry on tissue biopsy is required on most recent pathologic specimen prior to protocol enrollment. Secondary testing for H. pylori with stool and/or urea breath tests and/or serum antigen is strongly recommended. Testing for the MALT1 translocation (t11:18) is strongly recommended if tissue for testing is available.
* Female patients with childbearing potential must have a negative serum or urine pregnancy test (βhCG) within 1 week of RT administration or have a documented pregnancy test refusal.
* The effects of RT on the developing human fetus are harmful. For this reason and because RT used in this trial is known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of RT administration. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

  * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
  * History of hysterectomy or bilateral salpingo-oophorectomy.
  * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
  * History of bilateral tubal ligation or another surgical sterilization procedure.
* Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of RT administration, and 4 months after completion of RT administration.
* Ability to understand and the willingness to sign a written informed consent document.
* Patients with bulky tumors (>7.5 cm) are allowed.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial

Exclusion Criteria:

* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because RT is an agent with the potential for teratogenic or abortifacient effects.
* Patients with other lymphoma diagnoses other than marginal zone lymphoma.
* Patients with a history of radiation to the treated site, if re-treatment would exceed known gastric or surrounding critical structure (e.g., bowel, spinal cord) tolerance.
* Patients with active scleroderma under treatment are ineligible as prior studies have shown excessive toxicity in scleroderma patients treated with RT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Jillian Gunther, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org